CLINICAL TRIAL: NCT00000792
Title: A Pharmacologically Guided Phase I/II Study of Daily Orally Administered Synthetic Hypericin in HIV-Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: VIMRx Pharmaceuticals (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 258; 11235 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Administration, Oral; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — hypericin

INTERVENTIONS:
Drug: Hypericin

SUMMARY:
To determine the safety and tolerance of daily oral hypericin when given to achieve target trough levels within defined cohorts. To determine the responses of surrogate markers of HIV infection to daily oral hypericin.

It is not known whether daily oral dosing will produce a tolerable prolonged exposure to therapeutic levels of hypericin. Pharmacokinetic modeling studies have demonstrated that daily oral dosing should produce a trough level in a desired range without excessive peak levels.

DETAILED DESCRIPTION:
It is not known whether daily oral dosing will produce a tolerable prolonged exposure to therapeutic levels of hypericin. Pharmacokinetic modeling studies have demonstrated that daily oral dosing should produce a trough level in a desired range without excessive peak levels.

Cohorts of six patients each receive escalating doses of oral hypericin daily. Blood is sampled for peak and trough levels the second week of therapy. A computer modeling algorithm will use these levels to determine the appropriate dose needed for each patient to achieve the desired trough level. When three of six patients at a given dose have completed 3 weeks of therapy without evidence of dose-limiting toxicity, data will be reviewed to determine whether subsequent patients should be entered at the next higher dose. The MTD is defined as the dose level immediately below that at which grade 3 or worse toxicity is seen in three or more of six patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis.

Allowed:

* Rifabutin, ketoconazole, fluconazole, and acyclovir, provided the medication has been taken for at least 4 weeks prior to study entry without toxicity.
* Topical medications such as clotrimazole troches or nystatin suspension.

Patients must have:

* Documented HIV infection.
* CD4 count <= 350 cells/mm3.
* p24 antigen positive at >= 35 pcg/ml.
* No active opportunistic infection at study entry that would require curative or suppressive therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy for which systemic chemotherapy is required.
* Medically significant liver disease, orthostatic hypotension, hypertension, cardiac disease, seizure disorders, or lymphoma.
* Any medical condition that would interfere with evaluation of the patient.

Concurrent Medication:

Excluded:

* AZT, ddI, ddC, d4T, or any other antiretroviral medication.
* Interferon or other immunomodulating drugs.
* Cytotoxic chemotherapy.
* Foscarnet.
* Ganciclovir.
* Antimycobacterial drugs other than rifabutin.
* MAO inhibitors.
* Hypertension-inducing, nephrotoxic, or hepatotoxic drugs.
* Opiates.
* Drugs known to cause photosensitivity.

Prior Medication:

Excluded within 1 month prior to study entry:

* AZT, ddI, ddC, d4T, or any other antiretroviral medication.
* Interferon or other immunomodulating drugs.
* Cytotoxic chemotherapy.
* Preparations known to contain hypericin.

Excluded within 3 months prior to study entry:

* Ribavirin.
* Hyperforate (500 mg tablets or ampules for IV injection) manufactured by Kline.
* Psychotonin M Alcohol Extract manufactured by Steigerwald.
* Hypericin (40 mg vial) by VIMRx.

Excluded within 14 days prior to study entry:

* Foscarnet.
* Ganciclovir.
* Antimycobacterial drugs other than rifabutin.
* MAO inhibitors.
* Hypertension-inducing, nephrotoxic, or hepatotoxic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 1995-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentine FT, Study Chair; Crumpacker C, Study Chair
Locations (3):
- United States (3):
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - NY Univ. HIV/AIDS CRS, New York, New York

REFERENCES:
- [Background] Furner V, Bek M, Gold J. A Phase I/II unblinded dose ranging study of hypericin in HIV-positive subjects. Int Conf AIDS. 1991 Jun 16-21;7(2):199 (abstract no WB2071)
- [Background] Gulick RM, McAuliffe V, Holden-Wiltse J, Crumpacker C, Liebes L, Stein DS, Meehan P, Hussey S, Forcht J, Valentine FT. Phase I studies of hypericin, the active compound in St. John's Wort, as an antiretroviral agent in HIV-infected adults. AIDS Clinical Trials Group Protocols 150 and 258. Ann Intern Med. 1999 Mar 16;130(6):510-4. doi: 10.7326/0003-4819-130-6-199903160-00015. PMID 10075619